CLINICAL TRIAL: NCT03756103
Title: To Evaluate the Safety and Efficacy of SPH3127 on Treating Mild-moderate Essential Hypertension Patients: A Randomized, Double-Blinded, Dose-Exploration and Placebo-Controlled Study
Brief Title: Safety and Efficacy of SPH3127 on Treating Mild-moderate Essential Hypertension Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Collaborators: R&G Pharma Studies Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPH3127-201
Record Dates: First submitted 2018-11-16; First posted 2018-11-28 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Hypertension,Essential
Keywords: mild-moderate essential hypertension; SPH3127 tablet; renin inhibitor; efficacy; safety
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SPH3127 tablet Dose 1 (Experimental): Low-dose group
  Interventions: Drug: SPH3127 tablet Dose 1
- SPH3127 tablet Dose 2 (Experimental): Mid-dose group
  Interventions: Drug: SPH3127 tablet Dose 2
- SPH3127 tablet Dose 3 (Experimental): High-dose group
  Interventions: Drug: SPH3127 tablet Dose 3
- SPH3127 tablet Placebo (Placebo Comparator): Placebo Control group
  Interventions: Drug: SPH3127 tablet Placebo

INTERVENTIONS:
Drug: SPH3127 tablet Dose 1 — Oral SPH3127 tablet, a kind of renion inhibitor, 50 mg, once daily for 8 weeks.
  Other Names: renion inhibitor
  Arms: SPH3127 tablet Dose 1
Drug: SPH3127 tablet Dose 2 — Oral SPH3127 tablet, a kind of renion inhibitor, 100 mg, once daily for 8 weeks.
  Other Names: renion inhibitor
  Arms: SPH3127 tablet Dose 2
Drug: SPH3127 tablet Dose 3 — Oral SPH3127 tablet, a kind of renion inhibitor, 200 mg, once daily for 8 weeks.
  Other Names: renion inhibitor
  Arms: SPH3127 tablet Dose 3
Drug: SPH3127 tablet Placebo — Oral SPH3127 tablet placebo, once daily for 8 weeks.
  Other Names: renion inhibitor placebo
  Arms: SPH3127 tablet Placebo

SUMMARY:
SPH3127 tablet is a of renin inhibitor. It is expected to be a new drug for essential hypertension. This is a phase IIa trial which designed to evaluate its efficacy and safety on treating mild-moderate essential hypertension patients.

DETAILED DESCRIPTION:
This is a dose finding trial. Totally 120 mild-moderate essential hypertension patients will be enrolled. All the patients will be randomized (1:1:1:1) into four groups (SPH3127 50mg, SPH3127 100mg, SPH3127 200mg and placebo).

The trial has three phases: the screening phase, the leading phase and the treating phase.

The primary endpoints are the changes of DBP and SBP compared to the baseline after 8 weeks of treatment.

All the adverse events are required to be collected for safety analyzing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female who is 18 - 65 years old.
2. Subject who is meeting the diagnostic criteria of mild-moderate essential hypertension：mean seated Systolic Blood Pressure (SBP) (2~3 times average) ≥ 140 mmHg and ≤ 179 mmHg and mean seated Diastolic Blood Pressure (DBP) (2~3 times average)≥ 90 and ≤ 109 mmHg.
3. Laboratory testing should:

（1） GFR* ≥ 60mL/min （2） AST or ALT is less than 2 times upper limit of normal （3） Hemoglobin ≥ 90g/L （4） Serum potassium ≥ 3.5mmol/L and ≤ 5.5mmol/L *the conversion formulas for GFR* Male：GFR=186×（Scr)^-1.154×(age)^-0.203； Female：GFR=186×（Scr)^-1.154×(age)^-0.203×0.742； Serum creatinine(Scr) unit：µmol/L.

Exclusion Criteria:

1. Subject who is diagnosed as a secondary hypertension.
2. Subject who is suspected to be malignant hypertension, hypertensive emergency, hypertensive urgencies patients.
3. Subject who is at risk when the current anti-hypertensive therapy discontinued.
4. Subject who is suffered by chronic congestive heart failure (NYHA III and IV) or myocardial infarction within 6 months. Subject has had or is currently suffered by serious heart disease, such as unstable angina, cardiogenic shock, arrhythmia to that needs treatment, heart valve disease, hypertrophic cardiomyopathy, rheumatic heart disease, etc.
5. Subject who is suffered by severe cerebrovascular disease or shock within 6 months, such as hypertensive encephalopathy, cerebrovascular injury, cerebral hemorrhage, transient ischemic attack etc.
6. Subject who is suffered by severe or malignant retinopathy. The severe lesions is defined as retinal hemorrhage, micro aneurysm, cotton wool patches, hard exudate or a combination of these symptoms. The malignant lesions defined as the combination of severe retinopathy and optic disc edema.
7. Subject's medication compliance is not suitable for this trial (use of medication is <80% or >120% in the leading phase).
8. Subject whose work is associated with such condition as work at height, motor driver or operating dangerous machine etc.
9. Subject who is suffered by aorta-arteritis, large aneurysm or aortic dissection, severe subclavian artery stenosis in the past.
10. Subject who had a gastrointestinal surgery history that may significantly alter drug absorption, distribution, metabolism and excretion（For example: gastroectomy, gastroenteroanastomosis or enterectomy, gastric bypass, gastrointestinal anastomosis, gastrointestinal band surgery, etc.).
11. Subject who have drug allergy history and anaphylactic reaction.
12. Subject who is lactating, or is planning to pregnant within six months after the trial.
13. Subject whose diabetes is out of controlled. Defined as fasting blood-glucose is > 7.8 mmol/L or glycosylated hemoglobin is>7.5%.
14. Subject who has a history of malignant tumor.
15. Subject who has a history of mental disorders.
16. Subject who has abnormal thyroid function examination or abnormal urine protein check value in urine routine(Urine protein test result is a "+" is considered abnormal).
17. Subject who has participated clinical trials within past 3 months (as a subject).
18. Subject who is planning or in use of other non-antihypertensive drugs which may affect blood pressure（for example: Monoamine oxidase inhibitors, anesthetics, tricyclic and tetracyclic antidepressants, non-steroidal anti-inflammatory drugs, reproductive oral contraceptive pills, thyroid hormones, adrenocortical hormones, etc.).
19. Subject who is planning or in use of other antihypertensive drugs during the trial.
20. Subject who is alcohol abuse （adult male/female consume more than 25g of alcohol per day: 25g of alcohol is equivalent to 200 mL of yellow rice wine/wine (15 degrees), 780mL of beer (4 degrees), 62 mL of liquor (50 degrees)） or drug abuse.
21. Subject that investigators considered to be not suitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Chinese
Enrollment: 120 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Changes From Baseline in Seated Systolic Blood Pressure (SBP) and Seated Diastolic Blood Pressure (DBP) After 8 Weeks of Treatment. | Baseline to 54-58 days
  To compare the changes of SBP and DBP after 8 weeks of treatment between each group.

SECONDARY OUTCOMES:
Changes from Baseline in Seated SBP and DBP after 2, 4 and 6 Weeks of Treatment. | Baseline to 14±2, 28±2 and 42±2 days
  To compare the changes of seated SBP and DBP after 2, 4 and 6 weeks of treatment between each group.
Changes from Baseline in 24-hour Ambulatory Blood Pressure after 8 Weeks of Treatment. | Baseline to 54-58 days
  To compare the change from baseline in 24-hour ambulatory blood pressure in each group after 8 weeks of treatment.
Effectiveness Rate after 4 and 8 Weeks of Treatment. | Baseline to 28±2 and 56±2 days
  To compare the rates that SBP decreased more than 20 mmHg or DBP decreased more than 10 mmHg between each group after 4 and 8 weeks of treatment.
Hypertension Controlled Rates after 4 and 8 Weeks of Treatment. | Baseline to 28±2 and 56±2 days
  To compare the rates that seated SBP < 140 mmHg and DBP < 90 mmHg between each group after 4 and 8 weeks of treatment.
Changes from Baseline in Plasma Renin Activity (PRA) Following 2, 4, 6 and 8 Weeks of Treatment. | Baseline to 14±2, 28±2,42±2 and 56±2 days
  To compare the changes of plasma renin activity (PRA) in each group after 2, 4, 6 and 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, Doctor, Principal Investigator — Beijing Anzhen Hospital
Locations (10):
- China (10):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - Xiangya Hospital Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Second People's Hospital of Guangdong Province, Guangdong
  - Inner Mongolia Medical University Affiliated Hospital, Hohhot
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Xuzhou Central Hospital, Xuzhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang F, Liu L, Ruan H, Chen X, Zhang Y, Yu Z, Li Y, Guan Y, Wang J, Huang K, Yu S, Cao Y, Ding C, Chang L, Huang Y, Chen X, Lv Q, Ma C. A randomized, double-blind, placebo-controlled, phase IIa, clinical study on investigating the efficacy and safety of SPH3127 tablet in patients with essential hypertension. Hypertens Res. 2024 Jul;47(7):1925-1933. doi: 10.1038/s41440-024-01657-z. Epub 2024 Apr 17. PMID 38632457